CLINICAL TRIAL: NCT04053868
Title: Evaluating the Comparative Pharmacokinetics of Nicotine After Administration Via JUUL or Tobacco Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 19-28309; 2R01DA039264-04A1 (NIH)
Record Dates: First submitted 2019-08-09; First posted 2019-08-13 (Actual); Results first posted 2023-08-15 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Nicotine Administration & Dosage; E-cigarettes; Vaping; E-Liquid; Tobacco Smoking
MeSH Terms: conditions — Vaping; Tobacco Smoking | interventions — Tobacco Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Electronic Cigarette (Experimental): The participants will participate in a standardized vaping session using a JUUL E-cigarette device with a JUUL e-liquid pod.
  Interventions: Other: JUUL
- Tobacco Cigarette (Experimental): The participants will participate in a standardized smoking session using commercial tobacco cigarettes.
  Interventions: Other: Tobacco

INTERVENTIONS:
Other: JUUL — Electronic Cigarette
  Arms: Electronic Cigarette
Other: Tobacco — Tobacco Cigarette
  Arms: Tobacco Cigarette

SUMMARY:
This is an observational, crossover design that will examine the pharmacokinetics and pharmacodynamics of impact of smoking tobacco cigarettes or vaping the JUUL electronic cigarette.

DETAILED DESCRIPTION:
The goal of this study is to better understand the pharmacokinetic and pharmacodynamics responses produced by the JUUL e-cigarette, compared to tobacco cigarettes, in e-cigarette and tobacco cigarette smokers.

Specific Aim #1- To categorize the nicotine pharmacokinetic (PK) profile (maximum plasma concentration; time to maximum plasma concentration and area under the concentration-time curve) and compare when using the JUUL e-cigarette vs. a tobacco cigarette in a standardized manner.

Specific Aim #2- To categorize the nicotine PK profile (maximum plasma concentration; time to maximum plasma concentration and area under the concentration-time curve(AUC)) and compare when using the JUUL e-cigarette vs a tobacco cigarette when using the product ad libitum.

Specific Aim #3- To evaluate various outcomes following JUUL e-cigarette or tobacco cigarette use, both with standardized and ad lib use including: heart rate, plasma catecholamines, pulmonary function testing.

Specific Aim #4- To evaluate and compare the effects on craving, reward and satisfaction when using the JUUL e-cigarette vs. tobacco cigarette.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of medical history and limited physical examination, as described below:
* - Heart rate < 105 beats per minute (bpm)
* - - Considered out of range if both machine and manual readings are above/below these thresholds.
* - Systolic Blood Pressure < 160 and > 90*
* - Diastolic Blood Pressure < 100 and > 50*
* Age: >= 21 & <=70 years old
* Body Mass Index (BMI) <= 38.0 (at PI's discretion for higher BMI if no other concurrent health issues)
* Willingness to avoid combusted marijuana up to 48 hours before each study visit
* Nicotine strength of e-liquid of usual e-cigarette > 0 mg/ml
* Group 1 Experienced E-cigarette users
* - Current use of tobacco cigarettes (<5 cigarettes per day)
* - Current e-cigarette use at least 15 days out of the past 30 days of a non-mod e-cigarette
* Group 2 Primary Tobacco cigarette users:
* - Currently smoking >= 5 cigarettes per day
* - Current e-cigarette use must be < 5 times per month
* Saliva cotinine >=50 ng/ml or urine cotinine and/or NicAlert=6
* Must have a smart phone, computer, or tablet and internet access (for remote procedures)

Exclusion Criteria:

* Medical
* - Heart disease
* - Seizures
* - Cancer
* - Thyroid disease (okay if controlled with medication)
* - Diabetes
* - Hepatitis B or C or Liver disease
* - Glaucoma
* - Kidney disease or urinary retention
* - History of stroke
* - An ulcer in the past year
* - Active use of an inhaler for Asthma or Chronic Obstructive Pulmonary Disease (COPD)
* Psychiatric conditions
* - Current or past schizophrenia, and/or current or past bipolar disorder
* - Major depression, current or within the past year
* - Major personality disorder
* - Participants with current or past minor or moderate depression and/or anxiety disorders will be reviewed by the principal investigator (PI) and/or medical monitor and considered for inclusion
* - History of psychiatric hospitalizations are not exclusionary, but study participation will be determined as per PI's or medical monitor's approval
* Drug/Alcohol Dependence
* - Alcohol or illicit drug dependence within the past 12 months with the exception of those who have recently completed an alcohol/drug treatment program
* - Positive toxicology test for illicit drugs at the screening visit (Tetrahydrocannabinol (THC) & prescribed medications okay)
* - Opioid replacement therapy (including methadone, buprenorphine, or other)
* Psychiatric medications
* - Current regular use of any psychiatric medications is exclusionary, with the exception of Selective Serotonin Reuptake Inhibitor (SSRI) and serotonin-norepinephrine reuptake Inhibitor (SNRI) and current evaluation by the PI and/or medical monitor that the participant is otherwise healthy, stable, and able to participate
* Medications
* - Use of sympatholytic medications for cardiovascular conditions including hypertension (Example: beta and alpha-blockers)
* - Use of medications that are inducers of nicotine metabolizing enzyme CYP2A6 (Example: rifampicin, carbamazepine, phenobarbital, and other anticonvulsant drugs)
* - Concurrent use of nicotine-containing medications
* - Any stimulant medications (example: Adderall) generally given for attention deficit hyperactivity disorder (ADHD) treatment
* Use of Other Tobacco Products (OTP)
* - Any of the following products in combination more than 15 times in the past month
* - - smokeless tobacco (snus, oral snuff, chewing tobacco)
* - - pipes
* - - cigars, cigarillos, little cigars
* - - blunts, spliffs
* - - hookah
* Other/Misc. Chronic Health Conditions
* Fainting (within the last 30 days)
* Other "life threatening illnesses" as per PI's or medical monitor's discretion
* Pregnancy
* - Pregnancy (self-reported and urine pregnancy test)
* - Breastfeeding (determined by self-report)
* Concurrent participation in another clinical trial (at PI's discretion)
* Inability to read and write in English
* Planning to quit smoking or vaping within the next 60 days
* Recent onset or change (worsening) in cough, fever and/or abdominal symptoms (vomiting or pain) in the past two weeks
* Diagnosis of pneumonia in the past 3 months
* Uncomfortable with blood draws
* Known allergy to propylene glycol or vegetable glycerin

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal L Benowitz, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Current users of nicotine were recruited from the San Francisco Bay Area as healthy volunteers for this study.
Groups:
- EC Day 1/TC Day 2: Participants will be randomized into one of two groups. In this group, participants will be assigned to exclusively use a JUUL e-cigarette (EC) on Study Day 1. They will then crossover to exclusively use a tobacco cigarette (TC) on Study Day 2. They will vape the e-cigarette during a Standardized Session (one 3.5 second puff every 30 seconds for a total of 10 puffs) followed by a 2.5 hour abstinence period. They will then vape as they wish for 4 hours.
  Electronic cigarette (EC): JUUL e-cigarette device with a JUUL e-liquid pod.
  Tobacco cigarette (TC): Participants' usual brand of tobacco cigarettes.
- TC Day 1/EC Day 2: Participants will be randomized into one of two groups. In this group, participants will be assigned to exclusively use a tobacco cigarette (TC) on Study Day 1. They will then crossover to exclusively use a JUUL e-cigarette (EC) on Study Day 2. They will smoke the tobacco cigarette during a Standardized Session (one 3.5 second puff every 30 seconds for a total of 10 puffs) followed by a 2.5 hour abstinence period. They will then smoke as they wish for 4 hours.
  Electronic cigarette (EC): JUUL e-cigarette device with a JUUL e-liquid pod.
  Tobacco cigarette (TC): Participants' usual brand of tobacco cigarettes.
Period: Overall Study
Arm/Group | EC Day 1/TC Day 2 | TC Day 1/EC Day 2
Started | 10 | 7
Completed | 9 | 7
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: 17 participants met eligibility requirements and were willing to start the study. One participant only completed the e-cigarette arm of the study, so they were not included in the Outcome Measures analysis.
Groups:
- Overall Study: Participants will exclusively use a JUUL E-cigarette device with a JUUL e-liquid pod on one study day and then exclusively a traditional tobacco cigarette on the other study day. The order in which the products are used are randomized using a Latin Square design. All participants will use both products (e-cigarette and tobacco cigarette).
Arm/Group | Overall Study
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Mean Nicotine Exposure
Description: Plasma nicotine area under the concentrated time curve (AUC) (ng/ml*h)
Time Frame: Plasma collected at baseline (prior to any product use) and at 2, 5, 7, 10, 15, 30, 60, 90, and 118 minutes after end of standardized session.
Measure: Mean (Standard Deviation); unit: ng/ml*h
Groups:
- E-cigarette (JUUL): Participants will exclusively use a JUUL E-cigarette device with a JUUL e-liquid pod on one of the study days. They will vape the e-cigarette during a Standardized Session (one 3.5 second puff every 30 seconds for a total of 10 puffs) followed by a 2.5 hour abstinence period. They will then vape as they wish for 4 hours.
- Tobacco Cigarette: Participants will exclusively use a tobacco cigarette on one of the study days. They will smoke the cigarette during a Standardized Session (one 3.5 second puff every 30 seconds for a total of 10 puffs) followed by a 2.5 hour abstinence period. They will then smoke as they wish for 4 hours.
Arm/Group | E-cigarette (JUUL) | Tobacco Cigarette
Number analyzed (Participants) | 16 | 16
ng/ml*h | 4.6 (2.2) | 9.2 (5.8)

2. Secondary Outcome: Overall Mean Heart Rate Over Time
Description: Participant heart rate will be measured in beats per minute (bpm) at baseline (before any use of products) and at 2, 5, 7, 10, 15, 30, 45, 60, 75, 90, 100,and 118 minutes after the standardized sessions of e-cigarette and tobacco cigarette use. The mean of each time point will be averaged over time.
Time Frame: Up to 118 minutes after end of standardized session.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | E-cigarette (JUUL) | Tobacco Cigarette
Number analyzed (Participants) | 16 | 16
bpm | 69.4 (11.6) | 73.4 (13.1)

3. Secondary Outcome: Mean Systolic Blood Pressure Over Time
Description: Participant systolic blood pressure will be taken at Baseline (prior to use of any product) and at 5, 10, 15, 30, 45, 60, 75, 90, 100, and 118 minutes after the standardized sessions of e-cigarette and/or tobacco cigarette use on each arm. The mean of each time point will be averaged over time.
Time Frame: Up to 118 minutes after end of standardized session.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Tobacco Cigarette: Participants will exclusively use a tobacco cigarette on one of the study days. They will smoke the e-cigarette during a Standardized Session (one 3.5 second puff every 30 seconds for a total of 10 puffs) followed by a 2.5 hour abstinence period. They will then smoke as they wish for 4 hours.
Arm/Group | E-cigarette (JUUL) | Tobacco Cigarette
Number analyzed (Participants) | 16 | 16
mmHg | 123 (12.3) | 122 (11.8)

4. Secondary Outcome: Mean Diastolic Blood Pressure Over Time
Description: Participant diastolic blood pressure will be taken at Baseline (prior to use of any product) and at 5, 10, 15, 30, 45, 60, 75, 90, 100, and 118 minutes after the standardized session during e-cigarette and/or tobacco cigarette use on each arm. The mean of each time point will be averaged over time.
Time Frame: Up to 118 minutes after end of standardized session.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | E-cigarette (JUUL) | Tobacco Cigarette
Number analyzed (Participants) | 16 | 16
mmHg | 75.6 (12) | 76.9 (10.6)

5. Secondary Outcome: Mean Questionnaire of Smoking Urges (QSU) and Modified for E-cigarettes (mQSU) Score Over Time
Description: The QSU (Questionnaire of Smoking Urges) is a self-report survey, modified to replace "cigarette" with "e-cigarette" and "smoking" with "vaping" for use during both the tobacco cigarette and the E-cigarette Arm. This instrument is composed of 10 items; 5 items measuring desire/intention to smoke/vape with smoking/vaping perceived as rewarding (Factor 1), and 5 items measuring anticipation of relief from negative affect with an urgent desire to smoke/vape (Factor 2). Scores for each factor (1 and 2) range from 5-35 with higher scores indicating more severe craving. The mean and standard deviation will be reported.
Time Frame: Up to 118 minutes after end of standardized session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | E-cigarette (JUUL) | Tobacco Cigarette
Number analyzed (Participants) | 15 | 15
score on a scale
  Factor 1: desire/intention to smoke/vape with smoking/vaping perceived as rewarding | 20.9 (9.62) | 19.0 (9.96)
  Factor 2: anticipation of relief from negative affect with an urgent desire to smoke/vape | 13.5 (8.72) | 11.3 (8.28)

6. Secondary Outcome: Mean Minnesota Nicotine Withdrawal Scale (MNWS) Score Over Time
Description: The Minnesota Nicotine Withdrawal Scale is an 15-item self -report scale designed to measure the severity of craving and withdrawal symptoms experienced during smoking cessation. Each item is on a scale of 0 to 4 with 0=none to 4=Severe. The responses to each item are summed to produce a total withdrawal summary score with a possible range between 0 and 60, with higher scores indicating greater withdrawal symptom severity with greater scores indicating a higher level of severity in nicotine withdrawal symptoms overall. The mean and standard deviation will be reported.
Time Frame: Up to 118 minutes after end of standardized session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | E-cigarette (JUUL) | Tobacco Cigarette
Number analyzed (Participants) | 15 | 15
score on a scale | 12 (8.75) | 11 (8.03)

7. Secondary Outcome: Mean Cigarette Evaluation Scale (CES) and Modified for E-cigarettes (mCES) Score Over Time
Description: The CES is a self-report survey measuring smoking/vaping satisfaction, psychological reward, aversion, sensations, and craving reduction. This 12-item instrument has a total score range from 12 to 84, with higher scores indicating higher perception of the above factors. The mean and standard deviation will be reported.
Time Frame: Up to 240 minutes after end of standardized session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | E-cigarette (JUUL) | Tobacco Cigarette
Number analyzed (Participants) | 15 | 15
score on a scale | 49.5 (12.87) | 47.7 (14.18)

ADVERSE EVENTS:
Time Frame: Up to 1 month.
Groups:
- Electronic Cigarette: The participants will use a JUUL e-cigarette device with a JUUL e-liquid pod in a standardized vaping session consisting of one 3.5 second puff every 30 seconds for a total of 10 puffs. This will be followed by a 2.5 hour abstinence period. They will then use the JUUL e-cigarette as they wish (ad-lib use) for 4 hours.
- Tobacco Cigarette: The participants will use a tobacco cigarette in a standardized smoking session consisting of one 3.5 second puff every 30 seconds for a total of 10 puffs. This will be followed by a 2.5 hour abstinence period. They will then use the tobacco cigarette as they wish (ad-lib use) for 4 hours.
Arm/Group | Electronic Cigarette | Tobacco Cigarette
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 2/16 | 1/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Electronic Cigarette (N=16) | Tobacco Cigarette (N=16)
cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-06-07): https://cdn.clinicaltrials.gov/large-docs/68/NCT04053868/Prot_001.pdf
  • Statistical Analysis Plan (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT04053868/SAP_002.pdf
  • Informed Consent Form (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/68/NCT04053868/ICF_000.pdf